CLINICAL TRIAL: NCT02963636
Title: Proximity Work in Family Medicine Groups : the Impact of Pharmacists
Acronym: FMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: McGill University (Other); Fonds de la Recherche en Santé du Québec (Other Government); Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Line Guénette, Assistant professor, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 106238
Record Dates: First submitted 2016-02-17; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Health Services
Keywords: family medicine group; pharmacists; primary health care; pharmaceutical services; interprofessional relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmacist clinical intervention (Experimental): Patients exposed to the pharmacist intervention
  Interventions: Other: Pharmacist clinical intervention

INTERVENTIONS:
Other: Pharmacist clinical intervention — Pharmacists will make a clinical intervention with patients. They will review patient drug therapy already prescribed in their usual care. This includes a medication reconciliation, an assessment of drug related problems, an assessment of the regimen complexity and adherence to treatment. A care plan will be elaborated. Moreover, immediate and future interventions with the patient or other health professionals will be implemented and monitored. There will be no drug or devices tested, it is a human clinical intervention by a pharmacist.

SUMMARY:
The project objective is to evaluate the impact of the recent addition of pharmacists within family medicine groups (FMGs) on organizational and clinical parameters. The process by which changes occur and the level of pharmacists' activities will also be assessed. The ultimate goal of the project is the development of an accompanying guide to facilitate the work of the pharmacist in monitoring complex patients in primary care medical clinics.

ELIGIBILITY:
Inclusion Criteria:

* Willing to meet with the pharmacist and;
* Consuming drugs of four or more different pharmacological classes or having to take at least four doses per day and;
* aged 70 or over with at least two criteria of vulnerability or aged less than 70 with at least 3 criteria of vulnerability or had a recent loss of autonomy or in post- hospitalization with medication changes in the hospital.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of drug related problems | 3 to 6 months

SECONDARY OUTCOMES:
Regimen complexity | 3 to 6 months
  Medication regimen complexity index (MRCI)
Medication adherence | 3 to 6 months
  Proportion of days covered (PDC)
Quality of care provided by the clinical team (pharmacists, doctors, nurses, etc.) | 3 to 6 months
  Quality indicators (proposed by INESSS)

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS de la Capitale-Nationale, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No